CLINICAL TRIAL: NCT03075124
Title: Effect of External Counter Pulsation on Coronary Artery Disease (ECP-CAD)
Brief Title: Effect of External Counter Pulsation on Coronary Artery Disease
Acronym: ECP-CAD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eighth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Second Affiliated Hospital of Xi'an Jiaotong University (Other); Second Affiliated Hospital of Zhengzhou University (Other); Shanghai 10th People's Hospital (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Guifu Wu, Professor, MD, PhD, Eighth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYSU8001
Record Dates: First submitted 2017-02-28; First posted 2017-03-09 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Stable Chronic Angina; Coronary Artery Disease
Keywords: Coronary Artery Disease; external counter pulsation; major adverse cardiovascular events
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External Counter Pulsation group (Experimental): A standard ECP protocol involves 35 one-hour sessions (once per day, 5 days a week) and continuous for 7 weeks. ECP consists of three sets of pneumatic cuffs attached to each of the patient's legs at the calf and lower and upper thigh. The inflation of the cuffs is triggered by a computer, and timing of the inflation is based on the R wave of the electrocardiogram. The ECP therapist adjusts the inflation and deflation timing to provide optimal blood movement per a finger plethysmogram waveform reading.
  Interventions: Device: External Counter Pulsation
- Control group (No Intervention): Guideline-driven standard medical treatment

INTERVENTIONS:
Device: External Counter Pulsation — A standard ECP protocol involves 35 one-hour sessions (once per day, 5 days a week) and continuous for 7 weeks. ECP consists of three sets of pneumatic cuffs attached to each of the patient's legs at the calf and lower and upper thigh. The inflation of the cuffs is triggered by a computer, and timing of the inflation is based on the R wave of the electrocardiogram. The ECP therapist adjusts the inflation and deflation timing to provide optimal blood movement per a finger plethysmogram waveform reading.
  Arms: External Counter Pulsation group

SUMMARY:
Coronary artery disease (CAD) is prevalent worldwide and the leading cause of mortality of citizens, external counter pulsation (ECP) has been elucidated that it may release angina symptoms and improve the prognosis of CAD, however, no multi-center control clinical study has been reported for further recommendation. The aim of this study is to evaluate the effect of ECP on CAD. To address this assumption, investigators enroll participants with stable CAD and randomize them into control or ECP group, the ECP intervention will be carried out with a standard protocol which involves 35 one-hour sessions (5 days a week) for continuous 7 weeks, and the follow-up will last for 1 year. The primary endpoint is the 1-year composite cardiovascular events (CCE), secondary endpoints include frequency of angina pectoris, heart function, biomarkers of arteriosclerosis, exercise tolerance and endothelial function.

DETAILED DESCRIPTION:
CAD is the leading cause of non-tumor mortality in most countries, ECP is a non-invasive method which consists of three sets of pneumatic cuffs attached to each of the patient's legs at the calf and lower and upper thigh. The inflation of the cuffs is triggered by a computer, and timing of the inflation is based on the R wave of the electrocardiogram. The ECP therapist adjusts the inflation and deflation timing to provide optimal blood movement per a finger plethysmogram waveform reading. This produces a retrograde flow of blood in the aorta resulting in a diastolic augmentation of blood flow and also an increase in venous return, which leads to an improved coronary perfusion pressure during diastole. Cumulative evidences demonstrate that ECP can improve life quality and release refractory angina which is not optimally controlled despite optimal medical management and coronary revascularization in patients with CAD, though the previous multi-center control trial (PROBE-EECP) had been designed, no result about the effect of ECP on the prognosis of CAD has been reported. Thus, this study is designed to enroll 380 participants with stable CAD after evaluation of frequency of angina pectoris, heart function, biomarkers of arteriosclerosis, exercise tolerance and endothelial function, participants will be randomized into ECP intervention group or control group. All participants receive Guideline-driven standard medical treatment, ECP will be carried out with a standard protocol which involves 35 one-hour sessions (5 days a week) for continuous 7 weeks. Up to the end of ECP intervention, CCE will be follow up to 1 year, meanwhile, items as above will be retested for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of coronary artery disease;
* Signed informed consent.

Exclusion Criteria:

* Obvious aortic insufficiency;
* Aortic aneurysm;
* Aortic dissection;
* Coronary fistula or severe coronary aneurysm;
* Symptomatic Congestive heart failure;
* Valvular heart disease;
* Congenital heart diseases;
* Cardiomyopathies
* Cerebral hemorrhage within six months;
* Uncontrolled hypertension, defined as SBP≥180mmHg or DBP≥110mmHg;
* Lower limb infection;
* Deep venous thrombosis;
* Progressive malignancies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2018-06-08 (Estimated); Primary Completion 2019-05-28 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
composite cardiovascular events (CCE) | Change from Baseline at 1-year
  Sudden cardiac death, angina pectoris after infarction, recurrent myocardial infarction；rehospitalization rate

SECONDARY OUTCOMES:
Frequency of angina pectoris per week | Change from Baseline frequency at 1 year
  Frequency of angina pectoris
Dosage of Nitroglycerin use per week | Change from Baseline frequency and dosage at 1 year
  total dosage of nitroglycerin
6-minute walking distance | Change from Baseline distance at 1 year
  6-minute walking distance

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Tenth People's Hospital of Tongji University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University,, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: Undecided